CLINICAL TRIAL: NCT02430298
Title: Topical and Oral Melatonin for Preventing Concurrent Radiochemotherapy Induced Oral Mucositis and Xerostomia in Head and Neck Cancer Patients
Brief Title: Topical/Oral Melatonin for Preventing Concurrent Radiochemotherapy Induced Oral Mucositis/Xerostomia Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Collaborators: Ubon Ratchathani Cancer Hospital, Ubon Ratchathani (Unknown); General Drugs House Co.,LTD. (Other)
Responsible Party: Principal Investigator, Nutjaree Pratheepawanit Johns, Khon Kaen University, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MLT-MX
Record Dates: First submitted 2014-01-28; First posted 2015-04-30 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Matched placebo (Placebo Comparator): Drug: match placebo Drug: placebo suspension gargle for 2 minutes before radiation 15 minutes and placebo gelatin capsule taken orally after 21:00 hours each night throughout the study
  Interventions: Drug: Matched Placebo
- Melatonin (Active Comparator): Drug: Melatonin 20 mg/ 10 ml melatonin suspension gargle for 2 minutes before radiation 15 minutes and 20 mg melatonin gelatin capsule taken orally after 21:00 hours each night throughout the study
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — Drug: Melatonin 20 mg/ 10 ml melatonin suspension gargle for 2 minutes before radiation 15 minutes and 20 mg melatonin gelatin capsule taken orally after 21:00 hours each night throughout the study
  Other Names: 20 mg/10 ml melatonin suspensions; 20 mg melatonin gelatin capsule
  Arms: Melatonin
Drug: Matched Placebo — Drug: Melatonin 20 mg/ 10 ml placebo suspension gargle for 2 minutes before radiation 15 minutes and 20 mg placebo gelatin capsule taken orally after 21:00 hours each night throughout the study
  Other Names: 20 mg/10 ml placebo suspensions; 20 mg placebo gelatin capsule
  Arms: Matched placebo

SUMMARY:
The study evaluates the effect of melatonin for preventing concurrent radiochemotherapy induced oral mucositis and xerostomia and improving quality of life in head and neck cancer patients. This is a randomized, double-blind, placebo controlled trial conducted in head and neck cancer patients. Mixed-block randomization is used to divide eligible patients into two groups: melatonin 40 mg or matched placebo. The patients are required to take the studied drugs 20 mg suspensions before radiation and 20 mg capsules at night (after 21.00 pm) on the first night of radiation and continue for 7 weeks. Standard treatment is Radiation 2 Gy 5 fraction/week not more than 7 weeks with Cisplatin chemotherapy base regimen according to standard hospital protocol. Study endpoints are level of mucositis (CTCAE scale, WHO scale and MTS scores), level of xerostomia (CTCAE scale, VAS), QOL (FACT-H&N), pain (VAS 0-10) and adverse event frequency.

ELIGIBILITY:
Inclusion Criteria:

* New diagnostic of head and neck cancer patient who need treatment with radiation involved with the oral cavity area.
* Never received radiotherapy or chemotherapy
* Karnofsky performance status > 70%
* Stopped smoking
* Able to eat and swallow medications
* Written informed consent

Exclusion Criteria:

* Melatonin allergy
* Active oral cavity inflammation scar
* Pregnancy
* Creatinine clearance < 30 ml/min
* Active periodontal disease
* Steroids or pain killer drugs used for oral cavity pain except NSAIDs for thromboembolism prevention
* Currently use benzydamine mouthwash

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Percentage of occurrence of mucositis level 3 or more by using the criteria of CTCAE version 4.0, World Health Organization scale and MTSscores | Time to event (occurence of mucositis level 3) during 7 weeks of treatment
  Participants will be followed for severity of mucositis during the treatment period of 7 weeks

SECONDARY OUTCOMES:
Percentage of occurrence of xerostomia level 2 or more by using the criteria of CTCAE version 4.0 and the Visual Analogue Scale | Time to event (occurence of mucositis level 3) during 7 weeks of treatment
  Participants will be followed for severity of xerostomia during the treatment period of 7 weeks
Quality of Life (FACT- H&N Version 4) | Change from baseline in Trial Outcome Index scores at 7th week

CONTACTS AND LOCATIONS:
Locations (1):
- Ubon Ratchathani Cancer Hospital, Ubon Ratchathani, Changwat Ubon Ratchathani, Thailand